CLINICAL TRIAL: NCT04663828
Title: UNification of Treatments and Interventions for TInnitus Patients - Randomized Clinical Trial (UNITI-RCT)
Acronym: UNITI-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNITI Consortium (Network)
Collaborators: University Hospital Regensburg (Other); University Hospital Virgen de las Nieves (Other); Hospital Clinico Universitario San Cecilio (Other); Charite University, Berlin, Germany (Other); National and Kapodistrian University of Athens (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNITI
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Hearing Aids; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Four different types of interventions will be included in the RCT. Two of them mainly target on the auditory aspects of tinnitus (hearing aid fitting and sound therapy), whereas the other two mainly target the CNS (Structured Counselling and Cognitive Behavioral Therapy).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Structured counseling (Other): Patients will receive a structured counseling therapy
  Interventions: Other: Structured counseling
- Hearing Aids (Other): Patients will receive hearing aids support
  Interventions: Device: Hearing aids
- Cognitive behavioral therapy (Other): Patients will receive cognitive behavioral therapy
  Interventions: Other: Cognitive behavioral therapy
- Sound therapy (Other): Patients will follow a sound therapy program
  Interventions: Other: Sound therapy
- Combination of sound therapy and cognitive behavioral therapy (Other): Patients will receive a combination of sound therapy and cognitive behavioral therapy
  Interventions: Other: Cognitive behavioral therapy; Other: Sound therapy
- Combination of hearing aids and cognitive behavioral therapy (Other): Patients will receive a combination of hearing aids and cognitive behavioral therapy
  Interventions: Device: Hearing aids; Other: Cognitive behavioral therapy
- Combination of hearing aids and structured counseling (Other): Patients will receive a combination of hearing aids and structured counseling
  Interventions: Other: Structured counseling; Device: Hearing aids
- Combination of structured counseling and sound therapy (Other): Patients will receive a combination of structured counseling and sound therapy
  Interventions: Other: Structured counseling; Other: Sound therapy
- Combination of hearing aids and sound therapy (Other): Patients will receive a combination of hearing and sound therapy
  Interventions: Device: Hearing aids; Other: Sound therapy
- Combination of cognitive behavioral therapy and sound therapy (Other): Patients will receive a combination of cognitive behavioral therapy and sound therapy
  Interventions: Other: Cognitive behavioral therapy; Other: Sound therapy

INTERVENTIONS:
Other: Structured counseling — Structured patient education and counselling is considered as providing information to patients in order to empower them to better manage their disorder
  Arms: Combination of hearing aids and structured counseling; Combination of structured counseling and sound therapy; Structured counseling
Device: Hearing aids — Hearing aids are considered medical devices and are recommended to patients with a certain degree of hearing loss. Hearing aids amplify environmental sounds.
  Arms: Combination of hearing aids and cognitive behavioral therapy; Combination of hearing aids and sound therapy; Combination of hearing aids and structured counseling; Hearing Aids
Other: Cognitive behavioral therapy — This is a structured intervention and consists of a several week program both with noise exposure and structured interviews and expert-patient as well as patient-patient interaction in groups
  Arms: Cognitive behavioral therapy; Combination of cognitive behavioral therapy and sound therapy; Combination of hearing aids and cognitive behavioral therapy; Combination of sound therapy and cognitive behavioral therapy
Other: Sound therapy — Several sounds and music are used for tinnitus disorder
  Arms: Combination of cognitive behavioral therapy and sound therapy; Combination of hearing aids and sound therapy; Combination of sound therapy and cognitive behavioral therapy; Combination of structured counseling and sound therapy; Sound therapy

SUMMARY:
The study includes a 12-week treatment trial for chronic tinnitus patients using 4 different types of interventions (hearing aids, sound therapy, structured counseling, cognitive behavioral therapy) either as a single treatment or a combination of two treatments. There are several aims of the study: compare 1) single vs. combined treatments, 2) single treatments vs. other treatments, 3) ear and brain based interventions, 4) analyzing data of the clinical trial in combination with other recorded data (genetic and proteomic data, audiology data) to develop in silico models of tinnitus and a decision support system with the aim to aid in treatment decisions. This randomized controlled trial is harmonized over five clinical centers in Europe with the aim to include 100 patients per center and is part of the UNITI-project (UNification of treatments and Interventions for TInnitus patients) funded by the European Union's Horizon 2020 programme (grant agreement number 848261).

DETAILED DESCRIPTION:
The study will be conducted as a randomized controlled trial (RCT), which investigates the effect of four different tinnitus therapy approaches applied over a time period of 12 weeks as a single or rather a combinatory treatment in 100 chronic tinnitus patients. The protocol of the RCT is harmonized over five clinical centers across Europe with each center responsible for study procedures (regulations with respect to CGP, GDPR etc.) themselves. Thus, the present protocol is for the Regensburg part of the study. Used therapies are - hearing aid (HA), sound therapy (ST), structured counseling (SC) and cognitive behavioral therapy for tinnitus (CBT4T). HA fitting will be conducted with CE-marked hearing aids from Signia Hearing Aids (Sivantos Pte. Ltd., Singapore, Republic of Singapore/ WSAudiology, Lynge, Denmark) with respect to patients hearing profile according to a standardized procedure. ST will be performed via a specifically developed mobile application (according to the European regulations for medical software (IEC 62304, IEC 82304)). Patients can select among 64 standardized or individualized (according to their tinnitus characteristics) sounds presented at a maximum loudness of 85 dB. A standardized SC protocol will be provided via a mobile application (preferably), URL-links, e-mail or in printed form over a 12-week treatment period including 12 chapters (one per week). CBT4T will be held on a weekly basis in groups not bigger than 6 patients á 1.5-2 hours. All interventions will be carried out by staff with corresponding expertise (e.g., audiologist or psychologists) or specially trained study assistants by these experts.

Prior to the start of the study, potential participants will be online pre-screened with respect to inclusion and exclusion criteria. If the potential candidates are appropriate for a participation, they will be invited for a first visit on-site for a detailed screening of inclusion and exclusion criteria, and of health-related, tinnitus-specific, audiological examinations and electrophysiological measurements (auditory brainstem response, auditory middle latency response). Based on their determined hearing profile the decision will be made, whether there is an indication for the application of a HA. Accordingly, the sample of patients will be stratified into two groups: patients with an HA indication and those without an indication. If such a HA indication does not exist, patients will alternatively receive ST. Within these two groups (hearing aid indication - yes or no), patients will be randomly allocated to the intervention arms consisting of single and combinational interventions.

Single therapy:

* HA (in the group stratified for hearing aids)
* ST
* SC
* CBT4T

Combinational therapy:

* HA + ST (in the group stratified for hearing aids)
* HA + SC (in the group stratified for hearing aids)
* HA + CBT4T (in the group stratified for hearing aids)
* ST + SC
* ST + CBT4T
* SC + CBT4T

Screening and baseline as well as treatment start can be performed on the same day. In this case relevant assessments are only performed once. In addition, blood samples can be obtained during screening, baseline or a separate visit before treatment begin. Blood sampling is voluntary and does not have influence on participation of the study. After the baseline visit the respective intervention will start (at latest 4 weeks after the baseline, otherwise baseline measurements will be repeated) and last for 12 weeks. During an interim assessment after 6 weeks of treatment participants have to complete health-related and tinnitus-specific questionnaires again plus additional assessments of adverse events. Interventions will end after 12 weeks with a repetition of measurements made during baseline and another evaluation of adverse events. A follow-up measurement is planned 9 months after the first visit (baseline measurement). Moreover, an additional voluntary follow-up assessment can be done 12 months after the first visit. Each visit will have a duration of approximately 2-3 hours. Our primary outcome will focus on changes in tinnitus distress measured via the Tinnitus Handicap Inventory (THI; (Newman et al., 1996)). Participants can choose to cancel their participation in the study at any point without reasons or any disadvantages except the missing treatment. Intervention for a single participant can be cancelled in the case of a significant deterioration of tinnitus symptoms. Slight worsening might be possible but expected to short-term. In case of worsening, participants receive support by trained medical and psychological experts. Prior to the start of the study, it will be registered in clinicaltrials.gov. For detailed information about the study procedure, interventions and used measurement please see the attached "UNITI - clinical investigation plan".

Sample A planned sample size of N = 100 patients in Regensburg will be recruited from the clinic and polyclinic for ear, nose and throat medicine as well as from the clinic and polyclinic for psychiatry and psychotherapy both part of the University of Regensburg. Additional recruitment strategies such as marketing via newspaper etc. are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Primary complaint tinnitus
2. Chronic tinnitus (for at least 6 months based on history)
3. Age 18-80 years
4. Ability to understand and consent to the research / ability to participate (hearing ability, intellectual capacity, no plans for sabbaticals or long-term holidays, no (plans for) pregnancy)
5. A score of >22 on the Montreal Cognitive Assessment (MoCa), i.e. adults without mild cognitive impairment
6. Ability and willingness to use the UNITI mobile applications on their smartphones
7. A score of ≥ 18 in the Tinnitus Handicap Inventory (THI) of Newman et al. (1996)
8. Willing to use a hearing aid (if indication)
9. If a drug therapy with psychoactive substances (e.g. antidepressants, anticonvulsants) exists at the beginning of the therapeutic intervention, it must have been stable for at least 30 days. The therapy should remain constant during the duration of the study, but a necessary change is not an exclusion criterion. Any change in medication is documented in the CRF.

Exclusion Criteria:

1. Objective tinnitus / heartbeat-synchronous tinnitus as primary complaint
2. Start of any other tinnitus related treatments, especially hearing aids, structured counseling, sound therapy (with special devices; expecting long term effects) or cognitive behavioral therapy in the last 3 months before the start of the study
3. Otosclerosis / acoustic neuroma or other relevant ear disorders with fluctuation hearing
4. Present acute infections (acute otitis media, otitis externa, acute sinusitis)
5. Meniere's disease or similar syndromes (but not vestibular migraine)
6. Serious internal, neurological or psychiatric conditions
7. Epilepsy or other CNS disorders (brain tumor, encephalitis)
8. Clinically relevant drug, medication or alcohol abuse up to 12 weeks before study start
9. Missing written informed consent
10. Severe hearing loss - inability to communicate properly in the course of the study
11. One deaf ear

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
The effects of interventions in tinnitus distress | Through study completion, an average of 22 months
  The primary outcome will cover the domain tinnitus distress. The total score in the Tinnitus Handicap Inventory (THI; Newman et al., (1996)) is defined as the primary outcome measure for tinnitus distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Tinnituszentrum Regensburg, Regensburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoisswohl S, Langguth B, Schecklmann M, Bernal-Robledano A, Boecking B, Cederroth CR, Chalanouli D, Cima R, Denys S, Dettling-Papargyris J, Escalera-Balsera A, Espinosa-Sanchez JM, Gallego-Martinez A, Giannopoulou E, Hidalgo-Lopez L, Hummel M, Kikidis D, Koller M, Lopez-Escamez JA, Marcrum SC, Markatos N, Martin-Lagos J, Martinez-Martinez M, Martinez-Martinez M, Ferron MM, Mazurek B, Mueller-Locatelli N, Neff P, Oppel K, Perez-Carpena P, Robles-Bolivar P, Rose M, Schiele T, Schiller A, Simoes J, Stark S, Staudinger S, Stege A, Verhaert N, Schlee W. Unification of Treatments and Interventions for Tinnitus Patients (UNITI): a study protocol for a multi-center randomized clinical trial. Trials. 2021 Dec 4;22(1):875. doi: 10.1186/s13063-021-05835-z. PMID 34863270
- [Background] Simoes JP, Schoisswohl S, Schlee W, Basso L, Bernal-Robledano A, Boecking B, Cima R, Denys S, Engelke M, Escalera-Balsera A, Gallego-Martinez A, Gallus S, Kikidis D, Lopez-Escamez JA, Marcrum SC, Markatos N, Martin-Lagos J, Martinez-Martinez M, Mazurek B, Vassou E, Jarach CM, Mueller-Locatelli N, Neff P, Niemann U, Omar HK, Puga C, Schleicher M, Unnikrishnan V, Perez-Carpena P, Pryss R, Robles-Bolivar P, Rose M, Schecklmann M, Schiele T, Schobel J, Spiliopoulou M, Stark S, Vogel C, Wunder N, Zachou Z, Langguth B. The statistical analysis plan for the unification of treatments and interventions for tinnitus patients randomized clinical trial (UNITI-RCT). Trials. 2023 Jul 24;24(1):472. doi: 10.1186/s13063-023-07303-2. PMID 37488627
- [Derived] Schoisswohl S, Basso L, Simoes J, Engelke M, Langguth B, Mazurek B, Lopez-Escamez JA, Kikidis D, Cima R, Bernal-Robledano A, Bocking B, Bulla J, Cederroth CR, Crump H, Denys S, Escalera-Balsera A, Gallego-Martinez A, Gallus S, Goedhart H, Hidalgo-Lopez L, Jarach CM, Kader H, Koller M, Lugo A, Marcrum SC, Markatos N, Martin-Lagos J, Martinez-Martinez M, Muller-Locatelli N, Neff P, Niemann U, Perez-Carpena P, Pryss R, Puga C, Robles-Bolivar P, Rose M, Schecklmann M, Schiele T, Schleicher M, Schobel J, Spiliopoulou M, Stark S, Staudinger S, Stege A, Todtli B, Trochidis I, Unnikrishnan V, Vassou E, Verhaert N, Vogel C, Zachou Z, Schlee W. Single versus combination treatment in tinnitus: an international, multicentre, parallel-arm, superiority, randomised controlled trial. Nat Commun. 2025 Nov 21;16(1):10510. doi: 10.1038/s41467-025-66165-1. PMID 41271763
- See also: Publication of study protocol — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-021-05835-z#article-info
- See also: Publication of Statistical Analysis Plan SAP — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-023-07303-2